CLINICAL TRIAL: NCT00504777
Title: An Open Label Study to Evaluate the Safety, and Effect on Treatment Response, of MabThera in Combination With Methotrexate in Patients With Active Rheumatoid Arthritis Who Have Had an Inadequate Response or Intolerance to One or More Anti-TNF Agents.
Brief Title: A Study of MabThera (Rituximab) in Combination With Methotrexate in Patients With Rheumatoid Arthritis Who Have Had an Inadequate Response to Anti-TNF Agents.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20798
Record Dates: First submitted 2007-07-19; First posted 2007-07-20 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab; Methotrexate

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]; Drug: Methotrexate

INTERVENTIONS:
Drug: rituximab [MabThera/Rituxan] — 1000mg iv on days 1 and 15
Drug: Methotrexate — 10-25mg/week po or parenteral

SUMMARY:
This single arm study will assess the safety and efficacy of MabThera in combination with methotrexate in patients with rheumatoid arthritis who have had an inadequate response or intolerance to one or more anti-TNF agents. Patients will receive MabThera 1000mg i.v. on days 1 and 15, and methotrexate (10-25mg/week p.o. or parenteral), together with methylprednisolone 100mg i.v. prior to infusion of MabThera. The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* active rheumatoid arthritis;
* receiving outpatient treatment;
* an inadequate response, or intolerance, to >=1 anti-TNF agent.

Exclusion Criteria:

* other rheumatic autoimmune disease or inflammatory joint disease;
* concurrent treatment with any anti-TNF-alpha therapy;
* joint or osseous surgery during 8 weeks prior to recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- Taiwan (6):
  - Changhua
  - Kaohsiung City
  - Taichung
  - Taipei
  - Taoyuan District
  - Tapei

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab + Methotrexate (MTX): Participants received rituximab 1000 milligrams (mg) intravenously (IV) and 100 mg methylprednisolone IV on Days 1 and 15. Participants were to be receiving background MTX (10-25 mg weekly, oral or parenteral dose).
Period: Overall Study
Arm/Group | Rituximab + Methotrexate (MTX)
Started | 36
Completed | 35
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: all participants who recieved any part of an infusion.
Groups:
- Rituximab + MTX: Participants received rituximab 1000 mg IV, and 100 mg methylprednisolone IV on Days 1 and 15. Participants were to be receiving background MTX (10-25 mg weekly, oral or parenteral dose).
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.72 (13.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity Score Based on 28-Joint Count (DAS28)
Description: DAS28 was calculated from the number of swollen joints, or swollen joint count (SJC) and tender joint count (TJC) using the 28 joints count, the erythrocyte sedimentation rate (ESR) (measured in millimeters per hour [mm/hr]), and Patient Global Assessment of Disease Activity (participant rated arthritis activity assessment) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity. A clinically significant improvement in DAS28 was a change of at least 1.2 units.
Time Frame: Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Rituximab + MTX: Participants received rituximab 1000 mg IV and 100 mg methylprednisolone IV on Days 1 and 15. Participants were to be receiving background MTX (10-25 mg weekly, oral or parenteral dose).
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 36
scores on a scale
  Baseline | 5.51 (1.05)
  Week 24 | 4.39 (1.21)
  Change from Baseline to Week 24 | -1.12 (1.19)
Statistical Analysis 1: Comparison: Rituximab + MTX; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) Response
Description: ACR20/50/70 response defined as greater than or equal to (≥)20 percent (%), 50%, or 70% improvement, respectively, in TJC and SJC, and ≥20%/50%/70% improvement in at least 3 of 5 remaining ACR core measures: Patient Assessment of Pain, Patient Global Assessment of Disease Activity, Physician Global Assessment of Disease Activity, self-assessed disability based on the Health Assessment Questionnaire-Disability Index (HAQ-DI), and C-Reactive Protein (CRP).
Time Frame: Week 24
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 36
percentage of participants
  ACR20 | 2.78
  ACR50 | 0
  ACR70 | 0

3. Secondary Outcome: Percentage of Participants Achieving a Response by European League Against Rheumatism (EULAR) Category
Description: Percentage of participants with a EULAR response at Week 24 based on a scale of good response, moderate response, or no response. The DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders have a change from baseline greater than (>)1.2 with DAS28 less than or equal to (≤)3.2; moderate responders have a change from baseline >1.2 with DAS28 >3.2 to ≤5.1 or change from baseline >0.6 to ≤1.2 with DAS28 ≤5.1; non-responders have a change from baseline ≤0.6 or change from baseline >0.6 and ≤1.2 with DAS28 >5.1.
Time Frame: Week 24
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 36
percentage of participants
  Good response | 0
  Moderate response | 58.33
  No response | 41.67

4. Secondary Outcome: Change From Baseline in HAQ-DI Score
Description: The Stanford HAQ-DI is a patient-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to 8 component sets: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Responses in each component set are scored from 0 (without any difficulty) to 3 (unable to do). The highest score recorded for any question in a category determines the score for the category, unless aids, devices, or help from another person is required. The HAQ-DI score is calculated as the sum of the category scores divided by the number of categories scored, giving a possible range of scores from 0 to 3. Scores of 0 to 1 are generally considered to represent "mild to moderate difficulty", 1 to 2 as "moderate to severe disability", and 2 to 3 as "severe to very severe disability".
Time Frame: Week 24
Population: ITT Population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Rituximab + MTX
Number analyzed (Participants) | 36
scores on a scale
  Baseline | 1.07 (0.69)
  Week 24 | 0.81 (0.65)
  Change from Baseline to Week 24 | -0.26 (0.52)
Statistical Analysis 1: Comparison: Rituximab + MTX; Test type: Superiority or Other; p = 0.0054, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Rituximab + MTX
Serious Adverse Events (participants affected / at risk) | 3/36
Other Adverse Events (participants affected / at risk) | 22/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + MTX (N=36)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + MTX (N=36)
Leukocytosis (Blood and lymphatic system disorders) | 1
Mononucleosis syndrome (Blood and lymphatic system disorders) | 1
Dizziness (Cardiac disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Oesophageal candidiasis (Gastrointestinal disorders) | 1
Peptic ulcer (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Oedema peripheral (General disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Respiratory tract infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 8
Alanine aminotransferase increased (Investigations) | 1
Blood pressure decreased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Weight increased (Investigations) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Joint dislocation (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Insomnia (Psychiatric disorders) | 1
Menorrhagia (Reproductive system and breast disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.